CLINICAL TRIAL: NCT05240534
Title: Using Smart Displays to Implement Evidence-Based eHealth System for Older Adults With Multiple Chronic Conditions (NHLBI)
Brief Title: ElderTree Via a Voice Activated Device for Managing Chronic Health Conditions (NHLBI)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-0984; A195000 (Other: UW Madison); Protocol Version 3/2/2023 (Other: UW Madison); 1R61HL151870-01A1 (NIH); 5R33HL151870 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Conditions, Multiple
Keywords: Voice-activated "smart" technology; Older adults
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (ET-Text) (Placebo Comparator): Participants will receive ElderTree on a laptop.
  Interventions: Behavioral: ET-Text (Laptop)
- Experimental group (ET-Voice) (Experimental): Participants will receive ElderTree on a smart system.
  Interventions: Behavioral: ET-Voice (Smart System)

INTERVENTIONS:
Behavioral: ET-Text (Laptop) — ElderTree (ET) is based on the extensively tested Comprehensive Health Enhancement Support System (CHESS). ET is a "walled garden" free of ads, with design features based on older users' feedback as well as best-practice principles such as uncluttered screens and large type. Like all CHESS systems, ET uses computers to deliver key elements of successful interventions: long duration, ongoing outreach, prompts, monitoring, cognitive reframing, action planning, problem solving, self-tailoring, and peer support. ET-Text arm will access ET on Laptop.
  Arms: Control group (ET-Text)
Behavioral: ET-Voice (Smart System) — ElderTree (ET) is based on the extensively tested Comprehensive Health Enhancement Support System (CHESS). ET is a "walled garden" free of ads, with design features based on older users' feedback as well as best-practice principles such as uncluttered screens and large type. Like all CHESS systems, ET uses computers to deliver key elements of successful interventions: long duration, ongoing outreach, prompts, monitoring, cognitive reframing, action planning, problem solving, self-tailoring, and peer support. ET-Voice arm will access ET on a smart speaker. Voice-activated devices can potentially be easy to use, even by those with limited dexterity or computer experience.
  Arms: Experimental group (ET-Voice)

SUMMARY:
Multiple chronic conditions (MCCs) are costly and pervasive among older adults. MCCs account for 90% of Medicare spending, and 65% of Medicare beneficiaries have 3 or more chronic conditions; 23% have 5 or more. MCCs are often addressed in primary care, where time pressures force a focus on medication and lab results rather than self-management skills. Patients often struggle with treatment adherence and the emotional and physical burdens of self-management and health tracking. Chronic conditions reduce quality of life (QOL) and increase loneliness, which exacerbate those conditions.

The primary purpose of this study is to investigate whether a voice-based platform is better for delivering an electronic health intervention to older adults than a text/typing-based platform. We have an evidence-based electronic health intervention (Elder Tree, ET) that has been shown to improve quality of life, physical and socio-emotional health outcomes for older adults with multiple chronic conditions when delivered via a text/typing-based system. The current project would test whether such patients would benefit even more if ET were delivered via a voice-based system (vs. the text-based system) because they would use it more consistently. ET is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥60 years old;
* Have medical record diagnoses of at least 5 chronic conditions of which at least 3 must come from the following: hypertension, hyperlipidemia, obesity, prediabetes or diabetes, or depression;
* Be willing to share medical record data about healthcare use (30-day hospital readmissions and ER, urgent care, primary care, and specialty care visits);
* Allow researchers to share information with the patient's primary care provider

Exclusion Criteria:

* Require an interpreter
* Report no current psychotic disorder that would prevent participation
* Have no acute medical problem requiring immediate hospitalization
* Not report impairments preventing use of a computer or tablet (e.g. blind, deaf)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in functional health as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 v2.1. | Baseline, 6, 12, 18 months
  Participant reported measure of overall health and level of physical disability. There are 4 questions with a possible score of 4-16. Lower scores indicate worse outcomes.
Change in pain interference as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 v2.1. | Baseline, 6, 12, 18 months
  Participant reported measure of pain interference, there are 4 questions, with a possible score of 4-20. Higher scores indicate worse outcomes.
Change in pain intensity as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 v2.1. | Baseline, 6, 12, 18 months
  Participant reported measure of pain intensity, this is a single question, with a possible score of 0 to 10. Higher scores indicate worse outcomes.
Change in fatigue as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 v2.1. | Baseline, 6, 12, 18 months
  Participant reported measure of fatigue, there are 4 questions, with a possible score of 4-20. Higher scores indicate worse outcomes.
Change in sleep as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 v2.1. | Baseline, 6, 12, 18 months
  Participant reported measure of sleep disturbance, there are 4 questions, with a possible score of 4-20. Higher scores indicate worse outcomes.
Change in anxiety as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 v2.1. | Baseline, 6, 12, 18 months
  Participant reported measure of anxiety, there are 4 questions, with a possible score of 4-20. Higher scores indicate worse outcomes.
Change in depression as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 v2.1. | Baseline, 6, 12, 18 months
  Participant reported measure of depression, there are 4 questions, with a possible score of 4-20. Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Change in overall ElderTree use across the 12-month intervention | up to 12 months
  Amount of ElderTree use will be calculated by number of logons in the ET portal.
Change in healthcare use (primary care, specialist, urgent care, emergency room visits, and 30-day readmissions | Baseline, 6, 12, 18 months
  Data will be collected from electronic health record.
Change in health distress | Baseline, 6, 12, 18 months
  Lorig Health Distress Scale is a self-reported measure. It has questions about how participant feel and how things have been during the past month. It is a 4 item scale. Each item can be score from 0-none of the time to 5- all the time. Higher scores corresponds to more amount of time the participant has been distressed about health (e.g.,discouraged, worried, fearful, frustrated by health problems).
Change in function and disability | Baseline, 6, 12, 18 months
  Late Life Function and Disability Instrument (FDI) evaluates self-reported difficulty a person has in performing activities of daily living tasks. There are 41 items with response options of "none," "a little," "some," "quite a lot," and "cannot do." An additional eight items for participants who use a walking device. Scores range from 1-5 with higher scores indicating higher levels of functioning.
Change in well-being | Baseline, 6, 12, 18 months
  The World Health Organization- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental well being. The WHO-5 consists of five statements, which respondents rate from 'All of the time = 5' to 'At no time = 0'. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Change in symptom distress | Baseline, 6, 12, 18 months
  General Symptom Distress Scale & Bayliss Disease Burden Scale is a 16-item which assesses the extent of distress caused by physical symptoms. The higher scores indicating more symptom distress or burden.
Change in falls | Baseline, 6, 12, 18 months
  The number of falls in the last 6 months
ElderTree ease of use | 6, 12, 18 months
  This is a 9 item scale created for the study to assess the ease of use of ElderTree. Participants rate items on a 4-point scale, with options ranging from not at all (1) to very much so (4), with higher scores indicating finding ElderTree useful.

OTHER OUTCOMES:
Change in NIH Toolbox Loneliness Survey scores | Baseline, 6, 12, 18 months
  NIH Toolbox Loneliness Survey is a self-report measure that assesses perceptions of loneliness. Participants rate items on a 5-point scale, with options ranging from never (1) to always (5). This creates a raw score, which is then converted to a t-score, with higher scores indicating greater levels of loneliness.
ElderTree usefulness | 6, 12, 18 months
  This is a 9 item scale created for the study to assess the usefulness of ElderTree. Participants rate items on a 4-point scale, with options ranging from not at all (1) to very much so (4), with higher scores indicating finding ElderTree useful.

CONTACTS AND LOCATIONS:
Overall Officials: David H Gustafson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gustafson DH Sr, Mares ML, Johnston DC, Curtin JJ, Pe-Romashko K, Landucci G. Comparison of Smart Display Versus Laptop Platforms for an eHealth Intervention to Improve Functional Health for Older Adults With Multiple Chronic Conditions: Protocol for a Randomized Clinical Trial. JMIR Res Protoc. 2025 Apr 3;14:e64449. doi: 10.2196/64449. PMID 40080672